CLINICAL TRIAL: NCT03431857
Title: Retrospective and Prospective, Multi Centre Study on T.E.S.S® V2 Shoulder System
Brief Title: Multi Centre Study on TESS V2 Shoulder System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.E13
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis Shoulder; Fracture; Rheumatoid Arthritis; Avascular Necrosis; Rotator Cuff Tear; Revision
Keywords: Shoulder arthroplasty; Medical device; Shoulder prosthesis; Performance
MeSH Terms: conditions — Fractures, Bone; Arthritis, Rheumatoid; Osteonecrosis; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- TESS V2 Prosthesis: Single study patient cohort, including 106 patients who meet the inclusion/exclusion criteria and who received the TESS V2 shoulder prosthesis.
  Interventions: Device: TESS V2

INTERVENTIONS:
Device: TESS V2 — Patients requiring the TESS V2 prosthesis.

SUMMARY:
This study is a Post Market Clinical Follow-up study to fulfill the post market surveillance requirements. The data collected from this study will serve the purpose of confirming safety and performance of the TESS Shoulder System.

DETAILED DESCRIPTION:
The objective of this retrospective and prospective, multicenter, non-controlled Post Market Clinical Follow-up study is to evaluate the mid-term (5-year) clinical performance of the TESS Version 2 Anatomic and Reverse prostheses in shoulder arthroplasty. The primary outcome is defined as the clinical performance determined using Constant Score. The secondary outcomes are the passive and active mobility, the radiographic evaluation, the complications (including dislocation and revisions/removals) and survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Except in special cases, the "anatomic" type is indicated for:

  * Centered osteoarthritis of the shoulder
  * Humeral head fractures
  * Rheumatoid arthritis (with intact rotator cuff)
  * Avascular necrosis of the humeral head
* Except in special cases, the "reversed" type is indicated for:

  * Offset osteoarthritis of the shoulder
  * Massive and non-repairable rotator cuff tears
  * Rheumatoid arthritis (with degenerative rotator cuff)
* Revision in cases of:

  * Replacement of an "anatomic" prosthesis with a "reversed" prosthesis
  * Conversion of a hemi-arthroplasty into a total arthroplasty
  * Increasing the size of the stem (length and/or diameter)
  * Replacing a glenoid prosthesis
  * Replacing a competitor's prosthesis
  * In rare cases, removing a "reversed" prosthesis and replacing it with an "anatomic" prosthesis
* Additional inclusion criteria include

  * Patient who read, understood study information and gave informed consent (oral or written depending on specific local regulatory requirements)
  * Willing to return for follow-up evaluations

Exclusion Criteria:

* Local or systemic infections.
* Severe muscular, neurological, or vascular deficiency of the affected joint.
* Bone destruction or poor bone quality liable to affect the stability of the implant (Paget's disease, osteoporosis, etc.)
* Cases where the corolla cannot be two-thirds covered with bone stock and including the stem/corolla junction.
* Any concomitant complaint likely to affect the functioning of the implant.
* Allergy to any of the implant components.
* Local bone tumors.
* Patient over 18 under law supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of Total Shoulder Arthroplasty (primary or revision) who receive the TESS V2 and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-10-20 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (2):
- Orthokliniek Waasland, Sint-Niklaas, Belgium
- Institut Calot, Berck, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TESS V2 Prosthesis
Started | 106
Completed | 52 (52 subjects have completed the study, and 50 had complete data (all pages of CRF visit are complete))
Not Completed | 54
Not completed — Death | 6
Not completed — Lost to Follow-up | 41
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Single study patient cohort, including 106 patients who meet the inclusion/exclusion criteria and who received the TESS V2 shoulder prosthesis.
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The gender of 2 patients (1.9% of participants) was unspecified in the CRF.
  Participants
    number analyzed (Participants) | 104
    Female | 74
    Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height cm [Mean (Standard Deviation); unit: cm] — Population: Height was not available for 4 of the patients.
  cm
    number analyzed (Participants) | 102
    (all) | 163.7 (7.6)
Weight kg [Mean (Standard Deviation); unit: Kg] — Population: Weight was not available for 2 of the patients.
  Kg
    number analyzed (Participants) | 104
    (all) | 75.9 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Constant Shoulder Score
Description: The Constant Murley score is a multi-item scale assessing the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (0-15 points), activities of daily living (0-20 points), strength (0-25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (0-40 points). The results are here reported as final score, which ranges from 0 to 100, with 0 representing the worst and 100 the best shoulder function.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 99 (pre-operative) and 50 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 99
score on a scale
  Pre-operative | 27.36 (13.95)
  5 years follow-up: number analyzed (Participants) | 50
  5 years follow-up | 63.5 (9.86)

2. Secondary Outcome: Active Anterior Elevation
Description: The active mobility is measured with 4 movements: active anterior elevation, active lateral elevation, external rotation elbow to body (RE 1) and external shoulder rotation in abduction at 90° (RE 2). Active anterior elevation measures the extent to which a patient can elevate the arm anteriorly and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 92 (pre-operative) and 50 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 92
degrees
  Pre-operative | 89.02 (36.3)
  5 years follow-up: number analyzed (Participants) | 50
  5 years follow-up | 131 (19.09)

3. Secondary Outcome: Active Lateral Elevation
Description: The active mobility is measured with 4 movements: active anterior elevation, active lateral elevation, external rotation elbow to body (RE 1) and external shoulder rotation in abduction at 90° (RE 2). Active lateral elevation measures the extent to which a patient can elevate the arm laterally and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 91 (pre-operative) and 50 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 91
degrees
  Pre-operative | 72.57 (40.17)
  5 years follow-up: number analyzed (Participants) | 50
  5 years follow-up | 105.70 (17.67)

4. Secondary Outcome: Active External Rotation RE1
Description: The active mobility is measured with 4 movements: active anterior elevation, active lateral elevation, external rotation elbow to body (RE 1) and external shoulder rotation in abduction at 90° (RE 2). Active external rotation RE1 measures the extent to which a patient can rotate the bent arm externally and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 96 (pre-operative) and 50 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 96
degrees
  Pre-operative | 22.45 (18.58)
  5 years follow-up: number analyzed (Participants) | 50
  5 years follow-up | 34.80 (18.54)

5. Secondary Outcome: Active External Rotation RE2
Description: The active mobility is measured with 4 movements: active anterior elevation, active lateral elevation, external rotation elbow to body (RE 1) and external shoulder rotation in abduction at 90° (RE 2). Active external rotation RE2 measures the extent to which a patient can rotate the arm externally from a position of 90° of abduction and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 76 (pre-operative) and 49 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 76
degrees
  Pre-operative | 28.22 (26.1)
  5 years follow-up: number analyzed (Participants) | 49
  5 years follow-up | 61.94 (17.22)

6. Secondary Outcome: Passive Elevation
Description: The passive mobility is measured with 2 movements: elevation and external rotation elbow to body (RE 1). Passive elevation measures the extent to which the arm of the patient can be passively elevated in the plane of the scapula and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 95 (pre-operative) and 50 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 95
degrees
  Pre-operative | 112.32 (27.40)
  5 years follow-up: number analyzed (Participants) | 50
  5 years follow-up | 140.90 (18.15)

7. Secondary Outcome: Passive External Rotation
Description: The passive mobility is measured with 2 movements: elevation and external rotation elbow to body (RE 1). Passive external rotation elbow to body (RE 1) measures the extent to which the bent arm of the patient can be passively rotated externally and is here reported in degrees.
Time Frame: Pre-operative, 5 years follow-up
Population: Number of cases for each time point: 95 (pre-operative) and 49 (5 years follow-up).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 95
degrees
  Pre-operative | 28.37 (18)
  5 years follow-up: number analyzed (Participants) | 49
  5 years follow-up | 43.47 (19.13)

8. Secondary Outcome: Radiographic Evaluation
Description: A complete radiographic evaluation (front view 3 rotations, lateral view) is completed pre-operatively. For the post-operative radiographic evaluations, the form is simplified and contains two options: "unchanged" or "changed" when compared to the preoperative x-ray, with presence of radiolucencies and/or notching. The number of "changed" radiographic evaluations per time point are here reported.
Time Frame: Immediate post-operative, 6 weeks follow-up, 6 months follow-up, 1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up.
Population: Number of radiographies analysed: 90 immediately post-operative, 83 at 6 weeks follow-up, 85 at 6 months follow-up, 75 at 1 year follow-up, 59 at 2 years follow-up, 36 at 3 years follow-up, 22 at 4 years follow-up, 44 at 5 years follow-up.
Measure: Number; unit: changed radiographies compared to pre-op
Units Other Than Participants: radiographies
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 90
Number analyzed (radiographies) | 90
changed radiographies compared to pre-op
  Immediate post-operative | 2
  6 weeks follow-up: number analyzed (Participants) | 83
  6 weeks follow-up: number analyzed (radiographies) | 83
  6 weeks follow-up | 6
  6 months follow-up: number analyzed (Participants) | 85
  6 months follow-up: number analyzed (radiographies) | 85
  6 months follow-up | 7
  1 year follow-up: number analyzed (Participants) | 75
  1 year follow-up: number analyzed (radiographies) | 75
  1 year follow-up | 7
  2 years follow-up: number analyzed (Participants) | 59
  2 years follow-up: number analyzed (radiographies) | 59
  2 years follow-up | 11
  3 years follow-up: number analyzed (Participants) | 36
  3 years follow-up: number analyzed (radiographies) | 36
  3 years follow-up | 5
  4 years follow-up: number analyzed (Participants) | 22
  4 years follow-up: number analyzed (radiographies) | 22
  4 years follow-up | 1
  5 years follow-up: number analyzed (Participants) | 44
  5 years follow-up: number analyzed (radiographies) | 44
  5 years follow-up | 12

9. Secondary Outcome: Survivorship
Description: The Kaplan-Meier method is used to report implant survivorship. This outcome measures survivorship of the implanted devices from the date of implantation to the date of revision or intended revision up to 5 years post-operatively.
Time Frame: 5 years follow-up
Population: Number of cases analyzed for each time point: 102 implanted devices (immediate post-operative) and 43 implanted devices (5 years follow-up).
Measure: Number (95% Confidence Interval); unit: Percentage of implanted devices
Units Other Than Participants: implanted devices
Arm/Group | TESS V2 Prosthesis
Number analyzed (Participants) | 43
Number analyzed (implanted devices) | 43
Percentage of implanted devices | 94.4 [89.7 to 99.4]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted up to 5 years after surgery, when the last follow-up was performed and patients completed the study.
Description: Adverse events were collected in an Adverse Event Form, which gathers information on the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome.
Arm/Group | TESS V2 Prosthesis
All-Cause Mortality (participants affected / at risk) | 5/106
Serious Adverse Events (participants affected / at risk) | 44/106
Other Adverse Events (participants affected / at risk) | 16/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TESS V2 Prosthesis (N=106)
Revision (Surgical and medical procedures) | 6 (6) — 4 due to dislocation, 1 due to glenoid loosening after a fall, 1 due to patient's dissatisfaction because of limited mobility.
Knee arthroplasty (Surgical and medical procedures) | 4 (5)
Lumbar surgery (Surgical and medical procedures) | 1 (1)
Shoulder surgery (Surgical and medical procedures) | 6 (6) — Other shoulder-related surgical procedures
Hip arthroplasty (Surgical and medical procedures) | 3 (3)
Hand surgery (Surgical and medical procedures) | 1 (1)
Elbow arthroplasty (Surgical and medical procedures) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) — Death occurred in 1 patient
Respiratory infection (Infections and infestations) | 4 (5)
Stroke (Cardiac disorders) | 2 (3) — Death occurred in 1 patient
Cardiac arrest (Cardiac disorders) | 2 (2) — Death occurred in 1 patient
Urinary disorder (Renal and urinary disorders) | 2 (2)
Kidney disorder (Renal and urinary disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Fracture thoracical vertebrae (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Death
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Surgery
Knee wound (Musculoskeletal and connective tissue disorders) | 1 (1) — Surgery
Pubis bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Conservative treatment
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Surgery
Shoulder fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Conservative treatment
Pseudoarthritis rhizomelic (Musculoskeletal and connective tissue disorders) | 1 (1) — Hospitalization, infiltrations
Neuropathy and athrosis of inferior limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Radius fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Surgery
Osteoporosis, fractures (Musculoskeletal and connective tissue disorders) | 1 (1)
Acromio-clavicular arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rachialgia and scapulalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cubital and Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) — Neurolysis
Humerocubital ostephytes (Musculoskeletal and connective tissue disorders) | 1 (1) — Neurolysis
Dementia + respiratory infection (General disorders) | 1 (1) — Death
Weakness (General disorders) | 1 (1) — Hospitalization
Stress incontinence (General disorders) | 1 (1) — Surgery
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vitrectomy (Eye disorders) | 2 (2)
Head wound (Skin and subcutaneous tissue disorders) | 1 (1)
Cement effraction (Surgical and medical procedures) | 1 (1) — Surgery
Parkinson (Nervous system disorders) | 1 (1)
Hyperalgic lumbosciatic (Nervous system disorders) | 1 (1) — Hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TESS V2 Prosthesis (N=106)
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Heterotopic ossification (Musculoskeletal and connective tissue disorders) | 1 (1)
Nerve injury (Nervous system disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Neck pain, paresthesia (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Due to fall
Respiratory infection (Infections and infestations) | 1 (1)
Biceps rupture (Musculoskeletal and connective tissue disorders) | 1 (1) — On previous tenodesis
Reflex sympathetic syndrom (Nervous system disorders) | 1 (1)
Postoperative inflammation suspected (Infections and infestations) | 1 (1) — Resolved with no further consequences
Acromion inflammation (Musculoskeletal and connective tissue disorders) | 1 (1)
Acromial fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Screw breakage (Surgical and medical procedures) | 1 (1) — During screwing of inferior screw, the screw touched the Fukuda retractor and broke. Screw was maintained in place, and no problem occurred further.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2012-05-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT03431857/Prot_000.pdf